CLINICAL TRIAL: NCT01005836
Title: Community Clinic Test of Youth Anxiety and Depression Study
Brief Title: Community Clinic Test of Youth Anxiety Treatment
Acronym: YADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, John Weisz, Professor and Primary Investigator, Harvard University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH057347 (NIH)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Anxiety; Depression
Keywords: Cognitive behavioral therapy; Anxiety treatment; Depression treatment; Child treatment; Usual care
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cognitive-behavioral therapy: Anxiety (Experimental): CBT for child anxiety. Coping Cat.
  Interventions: Behavioral: Cognitive behavioral therapy for youth anxiety
- Usual care: Anxiety (Other): Usual clinic care
  Interventions: Other: Usual clinic care
- Cognitive behavioral therapy: depression (Experimental): CBT for youth depression. The Primary and Secondary Control Enhancement Training protocol.
  Interventions: Behavioral: Cognitive behavioral treatment for youth depression
- Usual care: Depression (Other): Usual clinic care for depression
  Interventions: Other: Usual clinic care

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for youth anxiety
  Other Names: Coping Cat
  Arms: Cognitive-behavioral therapy: Anxiety
Other: Usual clinic care
  Arms: Usual care: Anxiety; Usual care: Depression
Behavioral: Cognitive behavioral treatment for youth depression
  Other Names: PASCET
  Arms: Cognitive behavioral therapy: depression

SUMMARY:
Structured, manualized treatments have been developed for numerous mental health problems and disorders among children and adolescents, and a number of these have shown strong beneficial effects in clinical trials. Such findings have led to proposals that the empirically supported treatments be used to improve outcomes of conventional clinic treatment, which some research suggests may not be very effective. But can these lab-tested treatments actually work in service-oriented clinics with referred youth? Available evidence cannot tell us, because the therapists, conditions, and clientele in the laboratory efficacy tests tend to differ so markedly from those of clinical practice. To assess the clinical potential of efficacy-tested treatments, we need effectiveness research that tests these treatments in the crucible of clinical practice. To help begin this process, the proposed research focuses on a specific treatment program for a specific cluster of disorders: Kendall's (1994) cognitive-behavioral "Coping Cat" program for child and adolescent anxiety disorders. The program has shown unusually positive effects across a series of clinical trials in the U.S. and Australia, but it has never been tested in real-world clinical conditions. The proposed study will test the effectiveness of the treatment with clinic-referred youth, treated in community clinics, with the treatment carried out by clinic staff therapists. Some 128 youth, aged 9-14, referred for anxiety and diagnosed with anxiety disorders, will be randomly assigned to receive either the usual treatment in the clinic, or the Kendall program, carried out by clinic staff who have been trained to proficiency. Therapists for the two treatment conditions will also be chosen randomly, from a pool of volunteers. Outcome assessment at immediate post-treatment, 1-year, and 2-year follow-ups, will test effects across many outcomes. It is hypothesized that outcomes for youths treated using the cognitive-behavioral treatment will be superior to those treated using usual care.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-IV anxiety or depressive disorder

Exclusion Criteria:

* Pervasive developmental disorder
* Psychotic disorder
* Mental retardation

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 1998-02; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Weisz, PhD, Principal Investigator — Harvard University

REFERENCES:
- [Result] Weisz JR, Southam-Gerow MA, Gordis EB, Connor-Smith JK, Chu BC, Langer DA, McLeod BD, Jensen-Doss A, Updegraff A, Weiss B. Cognitive-behavioral therapy versus usual clinical care for youth depression: an initial test of transportability to community clinics and clinicians. J Consult Clin Psychol. 2009 Jun;77(3):383-96. doi: 10.1037/a0013877. PMID 19485581
- [Derived] Southam-Gerow MA, Weisz JR, Chu BC, McLeod BD, Gordis EB, Connor-Smith JK. Does cognitive behavioral therapy for youth anxiety outperform usual care in community clinics? An initial effectiveness test. J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):1043-52. doi: 10.1016/j.jaac.2010.06.009. Epub 2010 Jul 31. PMID 20855049